CLINICAL TRIAL: NCT04927403
Title: A Prospective Observational Study in the Context of an Internal Medicine Clinic for Naturopathy and Integrative Medicine
Brief Title: Integrative Therapy of Chronic Diseases
Acronym: InteChron
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universität Duisburg-Essen (Other)
Collaborators: Sozialstiftung Bamberg (Other); Bavarian State Ministry of Health and Care (Other Government); Charite University, Berlin, Germany (Other); Kliniken Essen-Mitte (Other)
Responsible Party: Principal Investigator, Jost Langhorst, Prof. Dr. med., Universität Duisburg-Essen
Other Study IDs: 20068
Record Dates: First submitted 2021-04-13; First posted 2021-06-16 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Chronic Disease
Keywords: irritable bowel syndrome; ulcerative colitis; Crohn's disease; pain patients; rheumatism; fibromyalgia syndrome; integrative medicine; naturopathy; irritable bowel disease; chronic pain syndrome; complementary medicine; post Covid syndrome; oncological diseases; day clinic
MeSH Terms: conditions — Chronic Disease; Irritable Bowel Syndrome; Colitis, Ulcerative; Crohn Disease; Rheumatic Diseases; Fibromyalgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Chronic gastroenterological diseases - inpatient stay and day clinic: Irritable Bowel Syndrome, Crohn's disease, Ulcerative colitis
  Interventions: Other: multimodal integrative naturopathic therapy concept
- Chronic Pain patients - inpatient stay and day clinic: Chronic pain syndrome, Rheumatism, Fibromyalgia
  Interventions: Other: multimodal integrative naturopathic therapy concept
- Oncological diseases - day clinic: all kinds of oncological diseases
  Interventions: Other: multimodal integrative naturopathic therapy concept
- post Covid syndrome - inpatient stay and day clinic: post Covid sydrome
  Interventions: Other: multimodal integrative naturopathic therapy concept
- other diseases - day clinic: e.g. patients with cardiovascular diseases, chron. Pulmonary diseases, metabolic disorders and skin diseases, etc.
  Interventions: Other: multimodal integrative naturopathic therapy concept

INTERVENTIONS:
Other: multimodal integrative naturopathic therapy concept — Use of conventional medicine, naturopathic approaches and complementary medical therapy methods

SUMMARY:
The observational study aims to investigate the extent to which a two-week stay in an internal medicine clinic for integrative medicine and naturopathy results in an improvement of complaints, impairments, quality of life, anxiety/depressiveness, stress perception and well-being in chronic gastroenterological patients and chronic rheumatological/pain patients. In addition, previous experiences with complementary naturopathic procedures, expectations of treatment, perceived benefits and implementation of instructed techniques and procedures in everyday life will be investigated.

Since May 2021, patients with Post Covid-19 Syndrome have been treated as inpatients during a stay that usually lasts 14 days. Since January 2022 these patients are evaluated in the substudy "StaPoCo". Since 2022 Post Covid-19 Syndrome day clinic patients were also evaluated.

Sub-Study "Intestinal barrier dysfunction" - Gastroenterological patients who undergo routine gastroscopy and/or colonoscopy with confocal laser endomicroscopy (cLE) and tissue biopsies at the beginning of their inpatient stay are explicitly examined for the presence of a barrier disorder.

Since May 2021 patients can take part in the day clinic programme one day weekly for ten or eleven weeks. In this programme also patients with oncological disorders take part.

Starting in the fall of 2022, the integrative medicine/naturopathic day clinics at the Immanuel Hospital in Berlin and the Ev. Kliniken Essen-Mitte will be included in the evaluation.

DETAILED DESCRIPTION:
This prospective uncontrolled observational study will include a minimum of 600 patients over six months. In the evaluation of the day clinic, the goal is at least 300 (up to approx. 600) patients. Primary outcome is general quality of life (SF-12). Secondary outcomes are anxiety and depression (HADS), well-being/flourishing (Flourishing), stress perception (PSS-10), and disease activity and disease-specific quality of life. In chronic gastroenterological patients, a distinction is made between patients suffering from irritable bowel syndrome (IBS-SSS + IBS-QOL), ulcerative colitis modifed MAYO Score + IBDQ) and Crohn's disease (HBI+ IBDQ). MAYO score: The partial MAYO score is used in this study. This contains only the non-invasive components of the full MAYO score, endoscopic findings are not considered. For chronic rheumatologic/pain patients, a distinction is made between pain patients in general (PDI), rheumatism (DAS-28, RAID), and fibromyalgia syndrome (Fibromyalgia Symptom Questionnaire, PHQ-15, PHQ-4, FIQ). The German Pain Questionnaire/ Severity Grading according to von Korff is applied to each of the three diseases. In addition, sociodemographics (age, gender, educational level, employment status, family situation), previous course of the disease, previous experience with/application of complementary medicine and naturopathic procedures, expectations of complementary medicine and naturopathic procedures used in the clinic, assessment and satisfaction with inpatient therapy program and planned and realized application of learned procedures are considered.

Substudy "StaPoCo" - In the case of post-Covid-19 disease, the Brief Pain Inventory (BPI), the MFI-20 questionnaire, the EQ-5D-5L are evaluated in addition to the modified baseline questionnaire, which is based on socio-demographic data, Covid-19 history. The survey of patients takes place at admission, discharge and after 6 months. Post-COVID-19 autoantibody screening (1xserum), as well as T-cell activation assay (Elispot) for the identification of potentially reactivated latent pathogens, such as EBV, CMV, VZV, TB and NTM (1xCPDA) (by biovis Diagnostics), which are scientifically discussed as potential causes for post-viral fatigue symptomatology, should be performed as part of the routine blood collection at admission (baseline) and discharge for post-COVID-19 inpatient patients.

Sub-Study "Intestinal barrier dysfunction" - Gastroenterological patients who undergo routine gastroscopy and/or colonoscopy with confocal laser endomicroscopy (cLE) and tissue biopsies at the beginning of their inpatient stay are explicitly examined for the presence of a barrier disorder. Patient groups: Crohn's disease (MC), ulcerative colitis (CU), irritable bowel syndrome (IBS). With this sub-study, the barrier disorder (primary or secondary) detected in the context of routine care and the corresponding therapies are to be observed in the course. At timepoints week 0 and after the end therapy (week 12-24) following parameters were assessed: the serum marker I-FABP and tissue samples for immunohistochemistry and gene expression analyzes, as well as the determination of food allergen-specific IgG/igG4 antibodies.

In the day clinic program also patients with oncological diseases (questionnaires: QLQ-C30 and FBK-R23) will be asked. In some day clinic groups a group discussion of about 45-60 minutes is to take place at the end of the treatment. Participants of the respective course who agree to take part in the group discussion, will be asked to make additional comments on the attended programme by means of standardised questionnaires.

Some participants (20) are also asked to take part in an individual telephone interview 6 months after completion of the programme. In this interview, the course of the patient's illness and the effects of participation in the day clinic on the illness and the patient's lifestyle in the past months are to be determined in more detail. A special focus is on the independent continuation of health-promoting measures after the end of the day clinic participation and the evaluation of supporting factors and obstacles in the implementation of the learned contents and techniques of the programme. The patients are selected on the basis of socio-demographic and clinical characteristics with the aim of obtaining a sample that is as heterogeneous as possible. The survey of patients takes place at the beginning of the day clinic, at the end of the programme (week 10 or 11) and after 6 months after the treatment.

The German Pain Questionnaire/ Severity Grading according to von Korff is applied to each of the three diseases. In addition, sociodemographics (age, gender, educational level, employment status, family situation), previous course of the disease, previous experience with/application of complementary medicine and naturopathic procedures, expectations of complementary medicine and naturopathic procedures used in the clinic, assessment and satisfaction with inpatient therapy program and planned and realized application of learned procedures are considered.

Starting in the fall of 2022, the integrative medicine/naturopathic day clinics at the Immanuel Hospital in Berlin and the Ev. Kliniken Essen-Mitte will be included in the evaluation. Since other patient groups are treated in Essen and Berlin (e.g., patients with cardiovascular diseases, chron. Pulmonary diseases, metabolic disorders and skin diseases, etc.), an additional questionnaire package was created for the indication group "Other diseases", in which the disease-specific symptoms are recorded using the MYMOP questionnaire. For the indication group "Rheumatic diseases", a questionnaire (HAQ) was added.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age
* signed declaration of consent

Exclusion Criteria:

* Patients who have not reached the age of 18.
* Expected life expectancy < 6 months (oncology patients).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who are admitted to the Clinic for Integrative Medicine and Naturopathy for inpatient treatment and belong to the following patient groups can participate:
  chronic gastroenterological patients: irritable bowel syndrome, ulcerative colitis, Crohn's disease chronic pain patients: rheumatism, fibromyalgia syndrome, chronic pain syndrome post Covid-19 syndrome patients: post Covid-19 syndromes oncological patients: all kinds of oncological diseases (only day clinic treatment)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Generic quality of life | week 0
  SF-12, Short Form 36 Health Survey Questionnaire
Generic quality of life | week 2 (inpatient), week 10/11 (day clinic)
  SF-12, Short Form 36 Health Survey Questionnaire
Generic quality of life | week 24 (inpatient), week 34/35 (day clinic)
  SF-12, Short Form 36 Health Survey Questionnaire

SECONDARY OUTCOMES:
anxiety and depression | week 0
  Hospital Anxiety and Depression Scale (HADS), 14 items (7 each for depressive symptoms or symptoms of anxiety). The two summated scores of the summated scales HADS-A and HADS-D range between 0 and 21. high scores indicate depressivness and anxiety
anxiety and depression | week 2 (inpatient), week 10/11 (day clinic)
  Hospital Anxiety and Depression Scale (HADS), 14 items (7 each for depressive symptoms or symptoms of anxiety). The two summated scores of the summated scales HADS-A and HADS-D range between 0 and 21. high scores indicate depressivness and anxiety
anxiety and depression | week 24 (inpatient), week 34/35 (day clinic)
  Hospital Anxiety and Depression Scale (HADS), 14 items (7 each for depressive symptoms or symptoms of anxiety). The two summated scores of the summated scales HADS-A and HADS-D range between 0 and 21. high scores indicate depressivness and anxiety
sex | week 0
  identification of the gender
age | week 0
  age in years
job | week 0
  identification of the current job (questionnaire)
Educational level | week 0
  identification of the educational level (questionnaire)
Expectation of the treatment (questionnaire) | week 0
  patient's expectations regarding treatment
Use of complementary medicine/natural remedies (questionnaire) | week 0
  medication and naturopathic approaches
Course of the disease (questionnaire) | week 0
  diagnosis, treatment methods, medication
wellbeing/flourishing | week 0 (inpatient stay)
  Flourishing Scale (FS-D), total value of the scale vary between 8 (minimum) and 56 (maximum). A high value corresponds to a person with many psychological resources and strengths
wellbeing/flourishing | week 2 (inpatient stay)
  Flourishing Scale (FS-D), total value of the scale vary between 8 (minimum) and 56 (maximum). A high value corresponds to a person with many psychological resources and strengths
wellbeing/flourishing | week 24 (inpatient stay)
  Flourishing Scale (FS-D), total value of the scale vary between 8 (minimum) and 56 (maximum). A high value corresponds to a person with many psychological resources and strengths
Perceived stress | week 0
  Perceived Stress Scale (PSS), Rating on a five-step scale from 1 (=never) to 5 (=very often), high stress is assumed from a total score of 20 points
Perceived stress | week 2 (inpatient), week 10/11 (day clinic)
  Perceived Stress Scale (PSS), Rating on a five-step scale from 1 (=never) to 5 (=very often), high stress is assumed from a total score of 20 points
Perceived stress | week 24 (inpatient), week 34/35 (day clinic)
  Perceived Stress Scale (PSS), Rating on a five-step scale from 1 (=never) to 5 (=very often), high stress is assumed from a total score of 20 points
disease activity (irritable bowel syndrome) | week 0
  IBS-SSS: To assess or evaluate the severity of the disease; the questionnaire includes 5 dimensions assessed with a visual analog scale (VAS): Severity of abdominal pain, frequency of abdominal pain, severity of abdominal distension, dissatisfaction with bowel habits, and impairment of quality of life.
disease activity (irritable bowel syndrome) | week 2 (inpatient), week 10/11 (day clinic)
  IBS-SSS: To assess or evaluate the severity of the disease; the questionnaire includes 5 dimensions assessed with a visual analog scale (VAS): Severity of abdominal pain, frequency of abdominal pain, severity of abdominal distension, dissatisfaction with bowel habits, and impairment of quality of life.
disease activity (irritable bowel syndrome) | week 24 (inpatient), week 34/35 (day clinic)
  IBS-SSS: To assess or evaluate the severity of the disease; the questionnaire includes 5 dimensions assessed with a visual analog scale (VAS): Severity of abdominal pain, frequency of abdominal pain, severity of abdominal distension, dissatisfaction with bowel habits, and impairment of quality of life.
diseasespecific quality of life (irritable bowel syndrome) | week 0
  The Irritable Bowel Syndrome Quality of Life (IBS-QOL) ; these are 34 items that reflect the impact of IBS on everyday life (0-100 points).
diseasespecific quality of life (irritable bowel syndrome) | week 2 (inpatient), week 10/11 (day clinic)
  The Irritable Bowel Syndrome Quality of Life (IBS-QOL) ; these are 34 items that reflect the impact of IBS on everyday life (0-100 points).
diseasespecific quality of life (irritable bowel syndrome) | week 24 (inpatient), week 34/35 (day clinic)
  The Irritable Bowel Syndrome Quality of Life (IBS-QOL) ; these are 34 items that reflect the impact of IBS on everyday life (0-100 points).
Partial Mayo Score, disease activity (ulcerative colitis) | week 0
  The Partial Mayo Scoring Index consists of a few questions for the patient to answer, and one question for the physician to answer. The numerical results provide a score that represents an estimate of ulcerative colitis disease severity.
Partial Mayo Score, disease activity (ulcerative colitis) | week 2 (inpatient), week 10/11 (day clinic)
  The Partial Mayo Scoring Index consists of a few questions for the patient to answer, and one question for the physician to answer. The numerical results provide a score that represents an estimate of ulcerative colitis disease severity.
Partial Mayo Score, disease activity (ulcerative colitis) | week 24 (inpatient), week 34/35 (day clinic)
  The Partial Mayo Scoring Index consists of a few questions for the patient to answer, and one question for the physician to answer. The numerical results provide a score that represents an estimate of ulcerative colitis disease severity.
diseasespecific quality of life (ulcerative colitis) | week 0
  Inflammatory Bowel Disease Questionnaire (IBD-Q), Recording on 7-point Likert scale, high values mean good, low values a reduced quality of life (1=worst score, 7=best score)
diseasespecific quality of life (ulcerative colitis) | week 2 (inpatient), week 10/11 (day clinic)
  Inflammatory Bowel Disease Questionnaire (IBD-Q), Recording on 7-point Likert scale, high values mean good, low values a reduced quality of life (1=worst score, 7=best score)
diseasespecific quality of life (ulcerative colitis) | week 24 (inpatient), week 34/35 (day clinic)
  Inflammatory Bowel Disease Questionnaire (IBD-Q), Recording on 7-point Likert scale, high values mean good, low values a reduced quality of life (1=worst score, 7=best score)
disease activity (Crohn's disease) | week 0
  Harvey-Bradshaw Index - HBI is used to assess the degree of illness in individuals with Crohn's disease. The highest possible sum is 30 points and indicates a severe course of disease. A lower sum than 5 points indicates a clinical remission.
disease activity (Crohn's disease) | week 2 (inpatient), week 10/11 (day clinic)
  Harvey-Bradshaw Index - HBI is used to assess the degree of illness in individuals with Crohn's disease. The highest possible sum is 30 points and indicates a severe course of disease. A lower sum than 5 points indicates a clinical remission.
disease activity (Crohn's disease) | week 24 (inpatient), week 34/35 (day clinic)
  Harvey-Bradshaw Index - HBI is used to assess the degree of illness in individuals with Crohn's disease. The highest possible sum is 30 points and indicates a severe course of disease. A lower sum than 5 points indicates a clinical remission.
diseasespecific quality of life (Crohn's disease) | week 0
  Inflammatory Bowel Disease Questionnaire (IBD-Q), Recording on 7-point Likert scale, high values mean good, low values a reduced quality of life (1=worst score, 7=best score)
diseasespecific quality of life (Crohn's disease) | week 2 (inpatient), week 10/11 (day clinic)
  Inflammatory Bowel Disease Questionnaire (IBD-Q), Recording on 7-point Likert scale, high values mean good, low values a reduced quality of life (1=worst score, 7=best score)
diseasespecific quality of life (Crohn's disease) | week 24 (inpatient), week 34/35 (day clinic)
  Inflammatory Bowel Disease Questionnaire (IBD-Q), Recording on 7-point Likert scale, high values mean good, low values a reduced quality of life (1=worst score, 7=best score)
disease activity (pain patients) | week 0
  Dt. Schmerzfragebogen/ Schweregraduierung nach von Korff -The intensity of the pain is determined with the help of the severity grading according to von Korff. On an 11-step rating scale (0 = no pain to 10 = strongest pain imaginable), the current, average and greatest pain intensity in the past 4 weeks is recorded. In addition, the extent of pain-related, subjectively experienced impairment is recorded for the areas of everyday life, leisure activities and ability to work.
disease activity (pain patients) | week 2 (inpatient), week 10/11 (day clinic)
  Dt. Schmerzfragebogen/ Schweregraduierung nach von Korff -The intensity of the pain is determined with the help of the severity grading according to von Korff. On an 11-step rating scale (0 = no pain to 10 = strongest pain imaginable), the current, average and greatest pain intensity in the past 4 weeks is recorded. In addition, the extent of pain-related, subjectively experienced impairment is recorded for the areas of everyday life, leisure activities and ability to work.
disease activity (pain patients) | week 24 (inpatient), week 34/35 (day clinic)
  Dt. Schmerzfragebogen/ Schweregraduierung nach von Korff -The intensity of the pain is determined with the help of the severity grading according to von Korff. On an 11-step rating scale (0 = no pain to 10 = strongest pain imaginable), the current, average and greatest pain intensity in the past 4 weeks is recorded. In addition, the extent of pain-related, subjectively experienced impairment is recorded for the areas of everyday life, leisure activities and ability to work.
diseasespecific quality of life (pain patients) | week 0
  The Pain Disability Index (PDI) was developed specifically for patients with pain. The German-language translation (Dillmann et al., 1994), which is consistent with the original in terms of content and form, consists of seven items that assess the impact of pain on individual domains of life: family and domestic obligations, leisure activities, social activities, occupation, sexual life, self-care, and activities essential to life. For each area, the patient is asked to indicate on an eleven-point scale the extent to which he or she is impaired here by his or her pain.
diseasespecific quality of life (pain patients) | week 2 (inpatient), week 10/11 (day clinic)
  The Pain Disability Index (PDI) was developed specifically for patients with pain. The German-language translation (Dillmann et al., 1994), which is consistent with the original in terms of content and form, consists of seven items that assess the impact of pain on individual domains of life: family and domestic obligations, leisure activities, social activities, occupation, sexual life, self-care, and activities essential to life. For each area, the patient is asked to indicate on an eleven-point scale the extent to which he or she is impaired here by his or her pain.
diseasespecific quality of life (pain patients) | week 24 (inpatient), week 34/35 (day clinic)
  The Pain Disability Index (PDI) was developed specifically for patients with pain. The German-language translation (Dillmann et al., 1994), which is consistent with the original in terms of content and form, consists of seven items that assess the impact of pain on individual domains of life: family and domestic obligations, leisure activities, social activities, occupation, sexual life, self-care, and activities essential to life. For each area, the patient is asked to indicate on an eleven-point scale the extent to which he or she is impaired here by his or her pain.
disease activity (rheumatism) | week 0
  The DAS (Disease Activity Score) is a scoring system developed by the European League of Rheumatism (EULAR). With the DAS28, the disease activity of rheumatoid arthritis is recorded on the basis of 28 defined joints (finger, hand, large joints) and a score between 0 and 10 is determined.
disease activity (rheumatism) | week 2 (inpatient), week 10/11 (day clinic)
  The DAS (Disease Activity Score) is a scoring system developed by the European League of Rheumatism (EULAR). With the DAS28, the disease activity of rheumatoid arthritis is recorded on the basis of 28 defined joints (finger, hand, large joints) and a score between 0 and 10 is determined.
disease activity (rheumatism) | week 24 (inpatient), week 34/35 (day clinic)
  The DAS (Disease Activity Score) is a scoring system developed by the European League of Rheumatism (EULAR). With the DAS28, the disease activity of rheumatoid arthritis is recorded on the basis of 28 defined joints (finger, hand, large joints) and a score between 0 and 10 is determined.
diseasespecific quality of life (rheumatism) | week 0
  Rheumatoid Arthritis Impact of Disease (RAID): Rheumatoid Arthritis Symptom Burden Questionnaire. The current questionnaire contains numeric scales from 0 to 10 for the assessment of pain, sleep, fatigue/exhaustion, impaired functioning, psychological well-being, situational awareness, and physical well-being.
diseasespecific quality of life (rheumatism) | week 2 (inpatient), week 10/11 (day clinic)
  Rheumatoid Arthritis Impact of Disease (RAID): Rheumatoid Arthritis Symptom Burden Questionnaire. The current questionnaire contains numeric scales from 0 to 10 for the assessment of pain, sleep, fatigue/exhaustion, impaired functioning, psychological well-being, situational awareness, and physical well-being.
diseasespecific quality of life (rheumatism) | week 24 (inpatient), week 34/35 (day clinic)
  Rheumatoid Arthritis Impact of Disease (RAID): Rheumatoid Arthritis Symptom Burden Questionnaire. The current questionnaire contains numeric scales from 0 to 10 for the assessment of pain, sleep, fatigue/exhaustion, impaired functioning, psychological well-being, situational awareness, and physical well-being.
disease activity and diseasespecific quality of life (rheumatism) | week 0
  Dt. Schmerzfragebogen/ Schweregraduierung nach von Korff -The intensity of the pain is determined with the help of the severity grading according to von Korff. On an 11-step rating scale (0 = no pain to 10 = strongest pain imaginable), the current, average and greatest pain intensity in the past 4 weeks is recorded. In addition, the extent of pain-related, subjectively experienced impairment is recorded for the areas of everyday life, leisure activities and ability to work.
disease activity and diseasespecific quality of life (rheumatism) | week 2 (inpatient), week 10/11 (day clinic)
  Dt. Schmerzfragebogen/ Schweregraduierung nach von Korff -The intensity of the pain is determined with the help of the severity grading according to von Korff. On an 11-step rating scale (0 = no pain to 10 = strongest pain imaginable), the current, average and greatest pain intensity in the past 4 weeks is recorded. In addition, the extent of pain-related, subjectively experienced impairment is recorded for the areas of everyday life, leisure activities and ability to work.
disease activity and diseasespecific quality of life (rheumatism) | week 24 (inpatient), week 34/35 (day clinic)
  Dt. Schmerzfragebogen/ Schweregraduierung nach von Korff -The intensity of the pain is determined with the help of the severity grading according to von Korff. On an 11-step rating scale (0 = no pain to 10 = strongest pain imaginable), the current, average and greatest pain intensity in the past 4 weeks is recorded. In addition, the extent of pain-related, subjectively experienced impairment is recorded for the areas of everyday life, leisure activities and ability to work.
disease activity (fibromyalgia syndrome) | week 0
  Fibromyalgia Symptom Questionnaire (FSQ) captures the severity of key fibromyalgia syndrome symptoms and the presence of various pain points over time in four sections.
disease activity (fibromyalgia syndrome) | week 2 (inpatient), week 10/11 (day clinic)
  Fibromyalgia Symptom Questionnaire (FSQ) captures the severity of key fibromyalgia syndrome symptoms and the presence of various pain points over time in four sections.
disease activity (fibromyalgia syndrome) | week 24 (inpatient), week 34/35 (day clinic)
  Fibromyalgia Symptom Questionnaire (FSQ) captures the severity of key fibromyalgia syndrome symptoms and the presence of various pain points over time in four sections.
symptom severity (fibromyalgia syndrome) | week 0
  Patient Health Questionnaire 15 (PHQ-15) consists of 15 items in the area of somatoform and depressive disorders. The PHQ-15 is scored by forming a sum score across all items. Symptom severity is assessed by the total score: minimal, mild, moderate, or severe.
symptom severity (fibromyalgia syndrome) | week 2 (inpatient), week 10/11 (day clinic)
  Patient Health Questionnaire 15 (PHQ-15) consists of 15 items in the area of somatoform and depressive disorders. The PHQ-15 is scored by forming a sum score across all items. Symptom severity is assessed by the total score: minimal, mild, moderate, or severe.
symptom severity (fibromyalgia syndrome) | week 24 (inpatient), week 34/35 (day clinic)
  Patient Health Questionnaire 15 (PHQ-15) consists of 15 items in the area of somatoform and depressive disorders. The PHQ-15 is scored by forming a sum score across all items. Symptom severity is assessed by the total score: minimal, mild, moderate, or severe.
symptom severity - depression and anxiety (fibromyalgia syndrome) | week 0
  PHQ-4 captures the dimensions of depression and anxiety with 4 items; patients are asked to indicate how often certain complaints (e.g., little happiness, dejection, anxiety) occurred over the course of the past two weeks
symptom severity - depression and anxiety (fibromyalgia syndrome) | week 2 (inpatient), week 10/11 (day clinic)
  PHQ-4 captures the dimensions of depression and anxiety with 4 items; patients are asked to indicate how often certain complaints (e.g., little happiness, dejection, anxiety) occurred over the course of the past two weeks
symptom severity - depression and anxiety (fibromyalgia syndrome) | week 24 (inpatient), week 34/35 (day clinic)
  PHQ-4 captures the dimensions of depression and anxiety with 4 items; patients are asked to indicate how often certain complaints (e.g., little happiness, dejection, anxiety) occurred over the course of the past two weeks
diseasespecific quality of life (fibromyalgia syndrome) | week 0
  The Fibromyalgia Impact Questionnaire (FIQ) is an instrument that quantifies the general impact of fibromyalgia syndrome in many dimensions. For example, it assesses functional ability, pain levels, fatigue, and sleep disturbances in patients affected by FMS. The FIQ is presented on a scale of 0-100, with a lower number indicating better health. It is a sensitive tool for therapy evaluation in fibromyalgia.
diseasespecific quality of life (fibromyalgia syndrome) | week 2 (inpatient), week 10/11 (day clinic)
  The Fibromyalgia Impact Questionnaire (FIQ) is an instrument that quantifies the general impact of fibromyalgia syndrome in many dimensions. For example, it assesses functional ability, pain levels, fatigue, and sleep disturbances in patients affected by FMS. The FIQ is presented on a scale of 0-100, with a lower number indicating better health. It is a sensitive tool for therapy evaluation in fibromyalgia.
diseasespecific quality of life (fibromyalgia syndrome) | week 24 (inpatient), week 34/35 (day clinic)
  The Fibromyalgia Impact Questionnaire (FIQ) is an instrument that quantifies the general impact of fibromyalgia syndrome in many dimensions. For example, it assesses functional ability, pain levels, fatigue, and sleep disturbances in patients affected by FMS. The FIQ is presented on a scale of 0-100, with a lower number indicating better health. It is a sensitive tool for therapy evaluation in fibromyalgia.
EQ-5D-5L Five dimensions of quality of life | week 0
  Dt. This questionnaire assesses the state of health (mobility, self-care, general activities, pain/physical discomfort and anxiety/dejection) as well as general health status on a VAS of 0-100. The questionnaire assesses is used for Post-Covid-Patients.
EQ-5D-5L Five dimensions of quality of life | week 2 (inpatient), week 10/11 (day clinic)
  Dt. This questionnaire assesses the state of health (mobility, self-care, general activities, pain/physical discomfort and anxiety/dejection) as well as general health status on a VAS of 0-100. The questionnaire assesses is used for Post-Covid-Patients.
EQ-5D-5L Five dimensions of quality of life | week 24 (inpatient), week 34/35 (day clinic)
  This questionnaire assesses the state of health (mobility, self-care, general activities, pain/physical discomfort and anxiety/dejection) as well as general health status on a VAS of 0-100. The questionnaire assesses is used for Post-Covid-Patients.
Pain and impairment (post-covid-19) | week 0 (inpatient stay)
  Dt. Brief pain inventory (BPI). It is used for Post-Covid-Patients. This questionnaire asks about pain and impairments in everyday life that occur due to these
Pain and impairment (post-covid-19) | week 2 (inpatient stay)
  Dt. Brief pain inventory (BPI). It is used for Post-Covid-Patients. This questionnaire asks about pain and impairments in everyday life that occur due to these.
Pain and impairment (post-covid-19) | week 24 (inpatient stay)
  Dt. Brief pain inventory (BPI). It is used for Post-Covid-Patients. This questionnaire asks about pain and impairments in everyday life that occur due to these
Lactoferrin (chronic gastroenterological) | week 0 (inpatient stay)
  Determination of lactoferrin in the stool
Lactoferrin (chronic gastroenterological) | week 2 (inpatient stay)
  Determination of lactoferrin in the stool
Lactoferrin (chronic gastroenterological) | week 24 (inpatient stay)
  Determination of lactoferrin in the stool
Calprotectin (chronic gastroenterological) | week 0 (inpatient stay)
  Determination of calprotectin in the stool
Calprotectin (chronic gastroenterological) | week 2 (inpatient stay)
  Determination of calprotectinin the stool
Calprotectin (chronic gastroenterological) | week 24 (inpatient stay)
  Determination of calprotectin in the stool
PMN-Elastase (chronic gastroenterological) | week 0 (inpatient stay)
  Determination of PMN-Elastase in the stool
PMN-Elastase (chronic gastroenterological) | week 2 (inpatient stay)
  Determination of PMN-Elastasethe in the stool
PMN-Elastase (chronic gastroenterological) | week 24 (inpatient stay)
  Determination of PMN-Elastasethe in the stool
Humanes Beta-Defensin (hBD-2) (chronic gastroenterological) | week 0 (inpatient stay)
  Determination of Humanes Beta-Defensin (hBD-2) in the stool
Humanes Beta-Defensin (hBD-2) (chronic gastroenterological) | week 2 (inpatient stay)
  Determination of Humanes Beta-Defensin (hBD-2) in the stool
Humanes Beta-Defensin (hBD-2) (chronic gastroenterological) | week 24 (inpatient stay)
  Determination of Humanes Beta-Defensin (hBD-2) in the stool
Zonulin (chronic gastroenterological) | week 0 (inpatient stay)
  Determination of zonulin in the stool
Zonulin (chronic gastroenterological) | week 2 (inpatient stay)
  Determination of zonulin in the stool
Zonulin (chronic gastroenterological) | week 24 (inpatient stay)
  Determination of zonulin in the stool
Alpha-Antitrypsin (chronic gastroenterological) | week 0 (inpatient stay)
  Determination of Alpha-Antitrypsin in the stool
Alpha-Antitrypsin (chronic gastroenterological) | week 2 (inpatient stay)
  Determination of Alpha-Antitrypsin in the stool
Alpha-Antitrypsin (chronic gastroenterological) | week 24 (inpatient stay - follow-up)
  Determination of Alpha-Antitrypsin in the stool
CRP (C-reactive protein) | week 0 (inpatient stay)
  Determination of CRP in the blood
CRP (C-reactive protein) | week 2 (inpatient stay)
  Determination of CRP in the blood
BKS (blood cell sedimentation rate) | week 0 (inpatient stay)
  Determination of BKS in the blood
BKS (blood cell sedimentation rate) | week 2 (inpatient stay)
  Determination of BKS in the blood
I-FABP (chronic gastroenterological - substudy) | inpatient stay (baseline)
  intestinal fatty-acid binding protein (blood)
I-FABP (chronic gastroenterological - substudy) | inpatient stay (up to 24 weeks)
  intestinal fatty-acid binding protein (blood)
IgG/IgG4 (chronic gastroenterological - substudy) | inpatient stay (baseline)
  immunoglobuline-G (blood)
IgG/IgG4 (chronic gastroenterological - substudy) | inpatient stay (up to 24 weeks)
  immunoglobuline-G (blood)
IgE (chronic gastroenterological - substudy) | inpatient stay (baseline)
  immunoglobuline-E (blood)
IgE (chronic gastroenterological - substudy) | inpatient stay (up to 24 weeks)
  immunoglobuline-E (blood)
tissue samples (chronic gastroenterological - substudy) | inpatient stay (baseline)
  Immunochemistry and gene expression analysis
tissue samples (chronic gastroenterological - substudy) | inpatient stay (up to 24 weeks)
  Immunochemistry and gene expression analysis
diseasespecific quality of life (oncological patients) | week 0 (day clinic)
  QLQ-C30: The EORTC QLQ-C30 questionnaire contains 30 questions and assesses the quality of life of oncological patients multidimensionally via 10 subscales. There are a number of additional modules for the disease-specific assessment of oncology patients.
diseasespecific quality of life (oncological patients) | week 11 (day clinic)
  QLQ-C30: The EORTC QLQ-C30 questionnaire contains 30 questions and assesses the quality of life of oncological patients multidimensionally via 10 subscales. There are a number of additional modules for the disease-specific assessment of oncology patients.
diseasespecific quality of life (oncological patients) | week 36 (day clinic)
  QLQ-C30: The EORTC QLQ-C30 questionnaire contains 30 questions and assesses the quality of life of oncological patients multidimensionally via 10 subscales. There are a number of additional modules for the disease-specific assessment of oncology patients.
psychological burden (oncological patients) | week 0 (day clinic)
  FBK-R23: Questionnaire on the Burden of Cancer Patients, 23 items on psychological, somatic and social burden.
psychological burden (oncological patients) | week 11 (day clinic)
  FBK-R23: Questionnaire on the Burden of Cancer Patients, 23 items on psychological, somatic and social burden.
psychological burden (oncological patients) | week 36 (day clinic)
  FBK-R23: Questionnaire on the Burden of Cancer Patients, 23 items on psychological, somatic and social burden.
monitoring of the main complaints (other diseases) | week 0 (day clinic)
  MYMOP: Measure Yourself Medical Outcome Profile
monitoring of the main complaints (other diseases) | week 10 (day clinic)
  MYMOP: Measure Yourself Medical Outcome Profile
monitoring of the main complaints (other diseases) | week 36 (day clinic)
  MYMOP: Measure Yourself Medical Outcome Profile
Questionnaire to assess disability due to inflammatory rheumatic joint disease | week 0 (day clinic)
  HAQ: Health assessment questionnaire, The patient fills out this questionnaire himself, assessing his ability to perform the following activities in eight daily functional areas: Dressing, standing up, eating, walking, personal hygiene, handing objects, grasping, other activities.
Questionnaire to assess disability due to inflammatory rheumatic joint disease | week 10 (day clinic)
  HAQ: Health assessment questionnaire, The patient fills out this questionnaire himself, assessing his ability to perform the following activities in eight daily functional areas: Dressing, standing up, eating, walking, personal hygiene, handing objects, grasping, other activities.
Questionnaire to assess disability due to inflammatory rheumatic joint disease | week 36 (day clinic)
  HAQ: Health assessment questionnaire, The patient fills out this questionnaire himself, assessing his ability to perform the following activities in eight daily functional areas: Dressing, standing up, eating, walking, personal hygiene, handing objects, grasping, other activities.
Post-COVID autoantibody screening and T-cell activation assay (Elispot) of potentially reactivated latent pathogens | week 0 (inpatient stay)
  blood collection (substudy StaPoCo)
Post-COVID autoantibody screening and T-cell activation assay (Elispot) of potentially reactivated latent pathogens | week 2 (inpatient stay)
  blood collection (substudy StaPoCo)
Questionnaire to measure the severity of tiredness in fatiguing illnesses (Post-Covid-19 syndrome) | week 0 (day clinic)
  Chalder Fatigue Scale
Questionnaire to measure the severity of tiredness in fatiguing illnesses (Post-Covid-19 syndrome) | week 10 (day clinic)
  Chalder Fatigue Scale
Questionnaire to measure the severity of tiredness in fatiguing illnesses (Post-Covid-19 syndrome) | week 36 (day clinic)
  Chalder Fatigue Scale
PSQI - Questionnaire which assesses sleep quality and disturbances (Post-Covid-19 Syndrome) | week 0 (day clinic)
  PSQI Pittsburgh Sleep Quality Index
PSQI - Questionnaire which assesses sleep quality and disturbances (Post-Covid-19 Syndrome) | week 11 (day clinic)
  PSQI Pittsburgh Sleep Quality Index
PSQI - Questionnaire which assesses sleep quality and disturbances (Post-Covid-19 Syndrome) | week 36 (day clinic)
  PSQI Pittsburgh Sleep Quality Index
MFI-20 - Multidimensional Fatigue Inventory (Post-Covid-19 Syndrome, substudy StaPoCo) | week 0 (inpatient stay)
  20-items rated on a 5-point scale (1 = "yes, that is true" to 5 = "no, that is not true") designed to evaluate five dimensions of fatigue: general fatigue, physical fatigue, reduced motivation, reduced activity, and mental fatigue. Higher scores represent more fatigue.
MFI-20 - Multidimensional Fatigue Inventory (Post-Covid-19 Syndrome, substudy StaPoCo) | week 2 (inpatient stay)
  20-items rated on a 5-point scale (1 = "yes, that is true" to 5 = "no, that is not true") designed to evaluate five dimensions of fatigue: general fatigue, physical fatigue, reduced motivation, reduced activity, and mental fatigue. Higher scores represent more fatigue.
MFI-20 - Multidimensional Fatigue Inventory (Post-Covid-19 Syndrome, substudy StaPoCo) | week 24 (inpatient stay)
  20-items rated on a 5-point scale (1 = "yes, that is true" to 5 = "no, that is not true") designed to evaluate five dimensions of fatigue: general fatigue, physical fatigue, reduced motivation, reduced activity, and mental fatigue. Higher scores represent more fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Jost Langhorst, Prof., Principal Investigator — Sozialstiftung Bamberg, Klinik für Integrative Medizin und Naturheilkunde
Locations (3):
- Germany (3):
  - Sozialstiftung Bamberg, Klinik für Intergrative Medizin, Bamberg, Bavaria
  - Evang. Kliniken Essen-Mitte, Klinik für Naturheilkunde & Integrative Medizin, Essen
  - Charité Hochschulambulanz für Naturheilkunde am Immanuel Krankenhaus Berlin, Standort Berlin-Wannsee, Wannsee

IPD SHARING:
Plan to Share IPD: No